CLINICAL TRIAL: NCT01805921
Title: A Phase I Study to Assess Safety and Immunogenicity of a New Respiratory Syncytial Virus (RSV) Vaccine Based on the RSV Viral Proteins F, N and M2-1 Encoded by Simian Adenovirus (PanAd3-RSV) and Modified Vaccinia Virus Ankara (MVA-RSV)
Brief Title: RSV001 - A New Vaccine to Prevent Severe Viral Chest Infections.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ReiThera Srl (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RSV001; 2011-003589-34 (EudraCT Number)
Record Dates: First submitted 2013-03-05; First posted 2013-03-06 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Respiratory Syncytial Virus; RSV; Vaccine
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- Arm 1. Prime PanAd3-RSV (IM), boost MVA-RSV (IM) (Experimental): Group 1A. Low dose prime PanAd3-RSV given by intra-muscular injection (IM) - low dose boost MVA-RSV given by intra-muscular injection (IM). 2 volunteers, 18-50 years. Interval: 8 weeks.
  Group 1B. High dose prime PanAd3-RSV given by intra-muscular injection (IM) - high dose boost MVA-RSV given by intra-muscular injection (IM). 8 volunteers, 18-50 years. Interval: 8 weeks.
  Interventions: Biological: MVA-RSV given by intra-muscular injection (high dose); Biological: PanAd3-RSV given by intra-muscular injection (high dose); Biological: MVA-RSV given by intra-muscular injection (low dose); Biological: PanAd3-RSV given by intra-muscular injection (low dose)
- Arm 2. Prime PanAd3-RSV (IM), boost PanAd3-RSV (IM) (Experimental): Group 2A. Low dose prime PanAd3-RSV given by intra-muscular injection (IM) - low dose boost PanAd3-RSV given by intra-muscular injection (IM). 2 volunteers, 18-50 years. Interval: 4 weeks.
  Group 2B. High dose prime PanAd3-RSV given by intra-muscular injection (IM) - high dose boost PanAd3-RSV given by intra-muscular injection (IM). 8 volunteers, 18-50 years. Interval: 4 weeks.
  Interventions: Biological: PanAd3-RSV given by intra-muscular injection (high dose); Biological: PanAd3-RSV given by intra-muscular injection (low dose)
- Arm 3. Prime PanAd3-RSV (IN), boost MVA-RSV (IM) (Experimental): Group 3A. Low dose prime PanAd3-RSV given intra-nasally (IN) - low dose boost MVA-RSV given by intra-muscular injection (IM). 2 volunteers, 18-50 years. Interval: 8 weeks.
  Group 3B. High dose prime PanAd3-RSV given intra-nasally (IN) - high dose boost MVA-RSV given by intra-muscular injection (IM). 8 volunteers, 18-50 years. Interval: 8 weeks.
  Interventions: Biological: PanAd3-RSV given intra-nasally (high dose); Biological: MVA-RSV given by intra-muscular injection (high dose); Biological: PanAd3-RSV given intranasally (low dose); Biological: MVA-RSV given by intra-muscular injection (low dose)
- Arm 4. Prime PanAd3-RSV (IN), boost PanAd3-RSV (IM) (Experimental): Group 4A. Low dose prime PanAd3-RSV given intra-nasally (IN) - low dose boost PanAd3-RSV given by intra-muscular injection (IM). 2 volunteers, 18-50 years. Interval: 8 weeks.
  Group 4B. High dose prime PanAd3-RSV given intra-nasally (IN) - high dose boost PanAd3-RSV given by intra-muscular injection (IM). 8 volunteers, 18-50 years. Interval: 8 weeks.
  Interventions: Biological: PanAd3-RSV given intra-nasally (high dose); Biological: PanAd3-RSV given by intra-muscular injection (high dose); Biological: PanAd3-RSV given intranasally (low dose); Biological: PanAd3-RSV given by intra-muscular injection (low dose)
- Arm 5. No vaccine (No Intervention): Group 5. Non-vaccinated control group. 6 volunteers, 60-75 years.
- Arm 6. MVA-RSV (IM) (Experimental): Group 6. Single high dose MVA-RSV given by intra-muscular injection (IM). 6 volunteers, 60-75 years.
  Interventions: Biological: MVA-RSV given by intra-muscular injection (high dose)
- Arm 7. Prime PanAd3-RSV (IM), boost PanAd3-RSV (IM) (Experimental): Group 7. High dose prime PanAd3-RSV given by intra-muscular injection (IM) - high dose boost PanAd3-RSV given by intra-muscular injection (IM). 6 volunteers, 60-75 years. Interval: 4 weeks.
  Interventions: Biological: PanAd3-RSV given by intra-muscular injection (high dose)
- Arm 8. Prime PanAd3-RSV (IN), boost MVA-RSV (IM) (Experimental): Group 8. High dose prime PanAd3-RSV given intra-nasally - high dose boost MVA-RSV given by intra-muscular injection (IM). 6 volunteers, 60-75 years. Interval: 8 weeks.
  Interventions: Biological: PanAd3-RSV given intra-nasally (high dose); Biological: MVA-RSV given by intra-muscular injection (high dose)
- Arm 9. Prime PanAd3-RSV (IM), boost MVA-RSV (IM) (Experimental): Group 9. High dose prime PanAd3-RSV given by intra-muscular injection (IM) - high dose boost MVA-RSV given by intra-muscular injection (IM). 6 volunteers, 60-75 years. Interval: 8 weeks.
  Interventions: Biological: MVA-RSV given by intra-muscular injection (high dose); Biological: PanAd3-RSV given by intra-muscular injection (high dose)

INTERVENTIONS:
Biological: PanAd3-RSV given intra-nasally (high dose) — High dose = 5x10^10 vp
  Arms: Arm 3. Prime PanAd3-RSV (IN), boost MVA-RSV (IM); Arm 4. Prime PanAd3-RSV (IN), boost PanAd3-RSV (IM); Arm 8. Prime PanAd3-RSV (IN), boost MVA-RSV (IM)
Biological: MVA-RSV given by intra-muscular injection (high dose) — High dose = 1x10^8 pfu
  Arms: Arm 1. Prime PanAd3-RSV (IM), boost MVA-RSV (IM); Arm 3. Prime PanAd3-RSV (IN), boost MVA-RSV (IM); Arm 6. MVA-RSV (IM); Arm 8. Prime PanAd3-RSV (IN), boost MVA-RSV (IM); Arm 9. Prime PanAd3-RSV (IM), boost MVA-RSV (IM)
Biological: PanAd3-RSV given by intra-muscular injection (high dose) — High dose = 5x10^10 vp
  Arms: Arm 1. Prime PanAd3-RSV (IM), boost MVA-RSV (IM); Arm 2. Prime PanAd3-RSV (IM), boost PanAd3-RSV (IM); Arm 4. Prime PanAd3-RSV (IN), boost PanAd3-RSV (IM); Arm 7. Prime PanAd3-RSV (IM), boost PanAd3-RSV (IM); Arm 9. Prime PanAd3-RSV (IM), boost MVA-RSV (IM)
Biological: PanAd3-RSV given intranasally (low dose) — Low dose = 5x10^9 vp
  Arms: Arm 3. Prime PanAd3-RSV (IN), boost MVA-RSV (IM); Arm 4. Prime PanAd3-RSV (IN), boost PanAd3-RSV (IM)
Biological: MVA-RSV given by intra-muscular injection (low dose) — Low dose = 1x10^7 pfu
  Arms: Arm 1. Prime PanAd3-RSV (IM), boost MVA-RSV (IM); Arm 3. Prime PanAd3-RSV (IN), boost MVA-RSV (IM)
Biological: PanAd3-RSV given by intra-muscular injection (low dose) — Low dose = 5x10^9 vp
  Arms: Arm 1. Prime PanAd3-RSV (IM), boost MVA-RSV (IM); Arm 2. Prime PanAd3-RSV (IM), boost PanAd3-RSV (IM); Arm 4. Prime PanAd3-RSV (IN), boost PanAd3-RSV (IM)

SUMMARY:
In this study we are testing a new vaccine against Respiratory Syncytial Virus (RSV).

This virus can cause respiratory infections such as bronchiolitis and pneumonia. It affects all ages, but especially infants, adults with a suppressed immune system, and the elderly. RSV only infects humans and occurs in epidemics each winter. It is the single most common cause of severe respiratory illness in children.

There is no effective anti-viral medication to treat RSV infections. There is a monoclonal antibody, which can be given to 'at-risk' children given by injection on a monthly basis during winter to provide short term protection against infection, but it is only partially effective and prohibitively expensive. Currently, there is no licensed vaccine to prevent RSV infection and there remains a real need to develop a vaccine as a cost-effective method to save lives and reduce the cost of disease caused by RSV.

DETAILED DESCRIPTION:
We are testing two new RSV vaccines, given in different combinations and by different routes of administration. Each vaccine uses the same RSV proteins to stimulate immune responses. These proteins are the F (Fusion), N (Nucleocapsid) and M2-1 (Matrix) proteins. The F protein sits on the surface of the virus and is needed to infect human cells. Antibodies to this protein are an important mechanism to prevent infection. The N and M2-1 proteins are needed for viral replication and are targets of immune recognition.

The two vaccines in this study contain all three of these proteins. However, they are delivered into the body using different 'vectors', which are harmless carrier viruses. In this study, we have employed two different vectors:a simian adenoviruses (PanAd3) and Modified Vaccinia virus Ankara (MVA).

We administer these vaccines using a 'prime-boost' strategy, in which one of these vaccines is used to 'prime' the immune system, which is then 'boosted' 4 or 8 weeks later, depending on the groups, by administration of an alternative vaccine or the same vaccine given by a different route.

ELIGIBILITY:
Inclusion Criteria:

Participants must satisfy all of the following criteria to be considered eligible for the study:

* Willing and able to give informed consent for participation in the study
* Aged between 18 and 50 years (Groups 1-4) or aged 60-75 years (Groups 5-9)
* In good health as determined by

  * Medical history
  * Physical examination
  * Clinical judgment of the investigators
* Willing to use effective contraception

  * Females: The oral contraceptive pill, contraceptive implant or barrier methods from one month prior and for the duration of the study (Groups 1-4 only)
  * Males: Barrier contraception from V1 until 3 months after the last vaccination
* Able to attend the scheduled visits and to comply with all study procedures
* Willing to allow his or her General Practitioner and/or Consultant, if appropriate, to be notified of participation in the study
* Confirmation from GP that they are aware of the inclusion and exclusion criteria and are satisfied from their knowledge of the volunteer that they are suitable to enroll
* Willing to provide their National Insurance/Passport number for the purpose of TOPS registration

Exclusion Criteria:

The participant may not enter the study if any of the following apply:

* History of significant organ/system disease that could interfere with trial conduct or completion. This includes any history of significant disease in the following;

  * Cardiovascular disease including congenital heart disease, previous myocardial infarction, valvular heart disease (or history of rheumatic fever), previous bacterial endocarditis, history of cardiac surgery (including pacemaker insertion), personal or family history of cardiomyopathy or sudden adult death
  * Respiratory disease such as asthma (excluding childhood asthma not treated in adulthood) and chronic obstructive pulmonary disease
  * Endocrine disorders such as diabetes mellitus and Addison's disease
  * Significant renal or bladder disease, including history of renal calculi
  * Biliary tract disease
  * Gastro-intestinal disease such as inflammatory bowel disease, abdominal surgery within the last two years, coeliac disease and liver disease
  * Neurological disease such as seizures and myasthenia gravis
  * Metabolic disease such as glucose-6-phosphate dehydrogenase deficiency
  * Psychiatric illness requiring hospitalization or depression whose severity is deemed clinical significant by the Chief Investigator, Consultant or GP
  * Non-benign cancer, including squamous cell carcinoma, basal cell carcinoma of the skin and cervical carcinoma in situ
  * Clinically significant contact dermatitis
* Have any known or suspected impairment or alteration of immune function, resulting from, for example:

  * Congenital or acquired immunodeficiency
  * Human Immunodeficiency Virus infection or symptoms/signs suggestive of an HIV-associated condition
  * Autoimmune disease
  * Receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 12 months or long-term systemic corticosteroid therapy
  * Receipt of immunoglobulin or any blood product transfusion within 3 months of study start
* A vaccination history indicative of;

  * Planning to receive any vaccine other than the study vaccine within 4 weeks following vaccination
  * A history of anaphylaxis reaction to a vaccine
  * History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, e.g. Kathon
  * Previously having received a recombinant simian or human adenoviral vaccine
  * Previously having received a recombinant MVA vaccine
* Detection of any of the following at screening

  * IgA deficiency
  * Anti-HIV antibody
  * Hepatitis B surface antigen
  * Anti-HCV antibody
  * Any other significant abnormalities on screening investigations at the discretion of an Investigator
* Known or suspected drug and/or alcohol misuse (alcohol misuse defined as an intake exceeding 42 units per week)
* Nasal septal pathology including

  * Congenital deformities such as an abnormal septum or polyps
  * Previous cauterization, rhinoplasty or surgery of any kind
  * Recurrent epistaxis
* Scheduled procedures requiring general anaesthesia during the study
* Participation in another research study involving an investigational product in the past 12 weeks, or are planning to do so within the 20 weeks of this study
* Inability, in the opinion of the Investigator, to comply with all study requirements
* Female participants who are pregnant, lactating or planning pregnancy during the course of the study
* Has donated blood within 4 months before starting the trial, or is intending to donate blood during the trial and up to 12 weeks after completing the study
* Any other significant disease or disorder which, in the opinion of the Investigator, may

  * Put the participants at risk because of participation in the study
  * Influence the result of the study
  * Impair the participant's ability to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-05; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Safety | 52 Weeks
  The recording and assessment of local and systemic adverse events following administration of each vaccine dose;
  * Fever
  * Headache
  * Nausea and/or vomiting
  * Malaise
  * Myalgia
  * Arthralgia
  * Injection site adverse events (for IM administered vaccine); pain or tenderness, induration, redness and swelling
  * Nasal site adverse events (for IN administered vaccine); pain or tenderness, irritation and discharge
  * Blood parameters
  * Any unsolicited symptom(s) not listed above

SECONDARY OUTCOMES:
Immunogenicity | 52 weeks
  Immunological assays to study immune responses to each vaccine, including:
  * Serum antibody response to RSV F antigen
  * Serum antibody response capable of RSV neutralization
  * Quantification of circulating vaccine-induced B-cell secreting antibodies (IgA and IgG) against RSV F antigen
  * Quantification of circulating vaccine-induced T-cell responses against RSV antigens F, N and M2-1
  * Any further exploratory immunology to detect vaccine related immune responses

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Pollard, FRCPCH PhD, Principal Investigator — University of Oxford. Department of Paediatrics
Locations (1):
- Centre for Clinical Vaccinology & Tropical Medicine (CCVTM), Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Derived] Green CA, Scarselli E, Voysey M, Capone S, Vitelli A, Nicosia A, Cortese R, Thompson AJ, Sande CS, de Lara C, Klenerman P, Pollard AJ. Safety and immunogenicity of novel respiratory syncytial virus (RSV) vaccines based on the RSV viral proteins F, N and M2-1 encoded by simian adenovirus (PanAd3-RSV) and MVA (MVA-RSV); protocol for an open-label, dose-escalation, single-centre, phase 1 clinical trial in healthy adults. BMJ Open. 2015 Oct 28;5(10):e008748. doi: 10.1136/bmjopen-2015-008748. PMID 26510727
- [Derived] Green CA, Scarselli E, Sande CJ, Thompson AJ, de Lara CM, Taylor KS, Haworth K, Del Sorbo M, Angus B, Siani L, Di Marco S, Traboni C, Folgori A, Colloca S, Capone S, Vitelli A, Cortese R, Klenerman P, Nicosia A, Pollard AJ. Chimpanzee adenovirus- and MVA-vectored respiratory syncytial virus vaccine is safe and immunogenic in adults. Sci Transl Med. 2015 Aug 12;7(300):300ra126. doi: 10.1126/scitranslmed.aac5745. PMID 26268313
- See also: More study information will be available from the Oxford Vaccine Group website once recruitment opens — http://www.ovg.ox.ac.uk/recruiting-studies